CLINICAL TRIAL: NCT01757951
Title: Unimalleolar Versus Bimalleolar Fixation in Bi- or Trimalleolar Ankle Fracture - A Randomized Clinical Trial
Brief Title: Unimalleolar Versus Bimalleolar Fixation in Bi- or Trimalleolar Ankle Fracture
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Partly due to financial issues and changes in study staff work placements
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Harri Pakarinen, MD, PhD, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OYSnilkka-RCT4
Record Dates: First submitted 2012-12-21; First posted 2012-12-31 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Trauma
Keywords: Ankle; Fracture; medial malleolus; Osteosynthesis
MeSH Terms: conditions — Wounds and Injuries; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unimalleolar Fixation (Experimental): Medial malleolus is fixed first and after that ankle mortise stability is assessed using external-rotation stress test. If talocrural joint is stable after fixation of medial malleolus, the patient is randomized to unimalleolar fixation group and no fixation of the lateral side is performed.
  Interventions: Procedure: Unimalleolar fixation
- Bimalleolar Fixation (Active Comparator): Medial malleolus is fixed first and after that ankle mortise stability is assessed using external-rotation stress test. If talocrural joint is stable after fixation of medial malleolus, the patient is randomized to bimalleolar fixation group i.e. additional fixation of the lateral malleolus fracture is performed.
  Interventions: Procedure: Bimalleolar fixation

INTERVENTIONS:
Procedure: Unimalleolar fixation — Medial malleolus is fixed first and after that ankle mortise stability is assessed using external-rotation stress test. If talocrural joint is stable after fixation of medial malleolus, the patient is randomized to unimalleolar fixation group and no fixation of the lateral side is performed.
  Arms: Unimalleolar Fixation
Procedure: Bimalleolar fixation — Medial malleolus is fixed first and after that ankle mortise stability is assessed using external-rotation stress test. If talocrural joint is stable after fixation of medial malleolus, the patient is randomized to bimalleolar fixation group i.e. additional fixation of the lateral malleolus fracture is performed.
  Arms: Bimalleolar Fixation

SUMMARY:
A one third of all ankle fractures are bi- or trimalleolar. Traditionally these fractures are treated by both medial and lateral osteosynthesis, sometimes accompanied by osteosynthesis of the posterior malleolus. There is significant evidence that fractures of the lateral malleolus can be treated conservatively if the medial side is stable. However, there isn't a single study comparing standard bi- or trimalleolar fixation with only medial side osteosynthesis and postoperative immobilization with a cast.

ELIGIBILITY:
Inclusion Criteria:

* Weber B bi- or trimalleolar ankle fracture (fracture of the lateral and medial malleolus +/- posterior malleolus sized under 30% of the distal tibia joint line measured from the lateral projection of the standard ankle radiographs)
* Age: 16 years or older
* Voluntary
* Operated within 7 days of the trauma
* Able to walk unaided before the current trauma

Exclusion Criteria:

* Peripheral neuropathy
* Pilon fracture
* Bilateral ankle fracture
* Concomitant tibial fracture
* Pathological fracture
* Active infection around the ankle
* A previous ankle fracture on either side
* In trimalleolar fractures, posterior malleolus fracture sized over 30% of the distal tibia joint line measured from the lateral projection of the standard ankle radiographs
* Inadequate co-operation
* Permanent residence outside the catchment area of the study hospital

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2012-02; Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Olerud-Molander Ankle Score | 2 years
  A validated, condition-specific, patient-reported measure of ankle fracture symptoms. Range from 0 to 100 points, with higher scores indicating better function

SECONDARY OUTCOMES:
The Foot and Ankle Outcome Score (FAOS) | 2 years
  FAOS, 5 subscales from 0-100, with higher scores indicating better function
A 100 mm Visual Analogue Scale for function and pain (VAS) | 2 years
  Range from 0 to 100, with higher scores indicating more severe pain
The RAND 36-Item Health Survey for health-related quality-of-life (RAND-36) | 2 years
  8 subscales from 0-100, with higher scores indicating better health-related quality of life
Talocrural joint congruence | At two, four and 12 weeks, and at 2 years
  Medial clear space < 4 mm and ≤ 1 mm wider than the superior clear space as measured between the lateral border of the medial malleolus and the medial border of the talus at the level of the talar dome.
Fracture healing | 2 years
  Fracture union is considered complete when the fracture line disappeared and conversely, those fractures with a visible fracture line are deemed non-unions.

OTHER OUTCOMES:
Complications and Harms | At two, four and 12 weeks, and at 2 years
  Treatment related complications and harms (i.e. wound infection, re-operations, deep vein trombhosis, plaster sore, wound healing problems)

CONTACTS AND LOCATIONS:
Overall Officials: Harri J Pakarinen, MD, PhD, AP, Study Director — Pohjois-Pohjanmaan sairaanhoitopiiri
Locations (1):
- Oulu University Hospital, Oulu, Finland